CLINICAL TRIAL: NCT06864767
Title: Impact of Motor and Oral Motor Function on Quality of Life in Children With Type I Spinal Muscular Atrophy
Brief Title: Impact of Motor and Oral Motor Function on Quality of Life in Children With SMA
Status: Completed | Type: Observational
Sponsor: Zeynep HOŞBAY (Other)
Responsible Party: Sponsor-Investigator, Zeynep HOŞBAY, Prof, Biruni University
Organization: Biruni University (Other)
Other Study IDs: Oral Motor Functions in SMA
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Spinal Muscular Atrophy Type I
Keywords: Spinal Muscular Atrophy Type I; Oral Motor Function; Motor Function; Quality of Life
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Neuro-sensory Motor Developmental Assessment — The test used to assess children's development levels evaluates the child's development in six parameters: gross motor function, fine motor function, neurological status, infant movement patterns, postural development and sensory-motor function (tactile, proprioceptive, ocular and vestibular systems) on a scale of 1 to 5. High scores are interpreted as motor dysfunction.
Other: Functional Oral Intake Scale — It is a scale consisting of a total of 7 levels and two sections, developed by Crary et al. to indicate the functional oral intake of patients with dysphagia. A higher score indicates a better nutritional level.
Other: Behavioral Pediatrics Feeding Assessment Scale — The scale used to determine eating problems in children evaluates both the child's nutritional status and the parents' feelings about the child's nutritional status. It consists of 35 items in total and is scored from 1 to 5. High scores indicate problematic eating behaviors and habits.
Other: Pediatric Quality of Life Inventory — The PedsQL assesses health-related quality of life in children ages 2 to 18 years with chronic illnesses from both the child's and parents' perspectives. It consists of 25 items and 3 categories (About My Child's Neuromuscular Disease, Communication, About Our Family Resources). The Neuromuscular Module was used to assess the quality of life of the children in our study and was answered by the parents only. The scale is scored from 0 to 4, with higher scores indicating better quality of life.

SUMMARY:
The aim of this study is to investigate the impact of motor and oral motor functions on the quality of life in children aged 2-4 years diagnosed with Spinal Muscular Atrophy (SMA) Type I. In the study, the Neuro-Sensory-Motor Developmental Assessment (NSMDA) was used to evaluate motor functions, the Functional Oral Intake Scale (FOIS) to assess oral motor function, the Behavioral Pediatric Feeding Assessment Scale (BPFAS) to evaluate children's attitudes towards feeding, and the Pediatric Quality of Life Inventory (PedsQL) Neuromuscular Module to assess quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Spinal Muscular Atrophy Type I
* Being between the ages of 2-4
* Families volunteering to participate in the study

Exclusion Criteria:

* Accompanied by another chronic disease other than SMA
* The mother or father has a cognitive problem that prevents them from expressing themselves
* The mother or father is illiterate

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study was completed with 23 children between the ages of 2-4 who were followed up with the diagnosis of Spinal Muscular Atrophy (SMA) Type 1 and whose parents volunteered to participate in the study.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Neuro-sensory Motor Developmental Assessment | Once, beginning of the study
  The test used to assess children's development levels evaluates the child's development in six parameters: gross motor function, fine motor function, neurological status, infant movement patterns, postural development and sensory-motor function (tactile, proprioceptive, ocular and vestibular systems) on a scale of 1 to 5. High scores are interpreted as motor dysfunction.
Functional Oral Intake Scale | Once, beginning of the study
  It is a scale consisting of a total of 7 levels and two sections, developed by Crary et al. to indicate the functional oral intake of patients with dysphagia. A higher score indicates a better nutritional level.
Behavioral Pediatrics Feeding Assessment Scale | Once, beginning of the study
  The scale used to determine eating problems in children evaluates both the child's nutritional status and the parents' feelings about the child's nutritional status. It consists of 35 items in total and is scored from 1 to 5. High scores indicate problematic eating behaviors and habits.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory | Once, beginning of the study
  The PedsQL assesses health-related quality of life in children ages 2 to 18 years with chronic illnesses from both the child's and parents' perspectives. It consists of 25 items and 3 categories (About My Child's Neuromuscular Disease, Communication, About Our Family Resources). The Neuromuscular Module was used to assess the quality of life of the children in our study and was answered by the parents only. The scale is scored from 0 to 4, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No